CLINICAL TRIAL: NCT02564172
Title: Conus Medullaris Stimulation With 5 Columns Lead Versus Medical Treatment in Refractory Pudendal Neuralgia: a Randomized, Open, Controlled, Multicenter Trial.
Brief Title: Conus Medullaris Stimulation With 5 Columns Lead Versus Medical Treatment in Refractory Pudendal Neuralgia
Acronym: STIMCONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0075
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pudendal Neuralgia
MeSH Terms: conditions — Pudendal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CMS group (Experimental): Conus medullaris stimulation with pentapolar surgical lead plus optimal medical management.
  Interventions: Device: CMS group
- OMM group (Active Comparator): Optimal medical management alone.
  Interventions: Other: OMM group

INTERVENTIONS:
Device: CMS group — Conus medullaris stimulation with pentapolar surgical lead includes:
  * Pentapolar surgical lead implant ((TM)Penta lead from St Judes Medical ANS which is the medical device under study)
  * Test phase of 10 days according to HAS("Haute Autorité de Santé") recommendation
  * If test phase positive, the lead is kept and subcutaneous rechargeable generator is implanted.
  * If test phase negative, the lead is removed.
  Optimal medical management : Similarly to patients randomized in active comparator group, patients randomized in experimental group will also be prescribed optimized medical management (treatment for pain relief) under algologist control.
  (A decrease of the consumption of pain treatment should be observed if conus medullaris stimulation has a positive effect).
  Other Names: Conus medullaris stimulation with pentapolar lead plus optimal medical management.
  Arms: CMS group
Other: OMM group — Optimal Medical Management (treatment for pain relief) includes analgesics and/or antidepressant and/or antiepileptics.Usually, drugs for neuropathic pain are prescribed as follows:
  * at effective dose, and minimal effective dose on the basis of adverse events and contraindications
  * as alone treatment in first and second line, then combination treatment. All this depends on the patient, on her/his pain, on her/his previous treatment.
  Medical treatment prescription will reviewed by algologist at each clinical visit. It is not possible in this indication to establish a standardized treatment.
  Non drugs therapies (physiotherapy, psychobehavioral approaches…) will not be forbidden or contra-indicated.
  Other Names: Optimal Medical Management alone.
  Arms: OMM group

SUMMARY:
Pudendal neuralgia is a frequent diagnosis in pain clinics. This perineal pain has devastating effects on patient's quality of life. Today, 30% of patients are refractory to pain management and surgical procedure.

The neuropathic characteristics of the pain in these patients lead us to test the efficiency of spinal cord stimulation at conus medullaris level.

In our published preliminary study involving 27 patients with refractory pudendal neuralgia, we demonstrated that 74% of patients implanted with stimulation electrodes at the conus medullaris responded to stimulation.

The primary objective of the present trial is to assess through a randomized, parallel group design, the effectiveness of spinal cord stimulation at the conus medullaris using pentapolar surgical lead ((TM)Penta, St Jude medical ANS) versus medical treatment alone on sitting time in refractory pudendal neuralgia.

DETAILED DESCRIPTION:
In this national multicenter prospective open label trial, patients will be randomized 1:1 to experimental group (CMS group : Conus Medullaris Stimulation using pentapolar surgical lead, plus optimal medical management) or to control group (OMM group : optimal medical management alone) and followed for 12 months, in intention to treat.

42 patients suffering of refractory pudendal neuralgia will be included. Optimal medical management will be prescribed by algologists in both groups according to patient pain relief.

ELIGIBILITY:
PRE-SCREENING CRITERIA:

* Male or female aged 18 years or over
* Pudendal neuralgia according published Nantes criteria
* History of failure medical management : defined by HAS such as intractable pain after failure (by side effect, ineffective, or contraindication) at effective dose and combination of following treatment:

  * Pain treatment OMS analgesics Level I or II
  * Tricyclicantidepressant
  * Antiepileptics
  * Nerve block
  * Muscle relaxants
  * Physiotherapy
  * TENS (Transcutaneus electric nerve stimulation)
  * Psychobehavioral approach
* Failure of pudendal nerve decompression surgery performed more than 12 months ago
* Neuropathic pain according to criteria of the Neuropathic Pain Diagnostic Questionnaire (DN4).
* Subjects able of giving informed consent
* Affiliation with French social security system.
* Average or maximum pain experienced greater than or equal to 5/10 on a visual analogue scale

INCLUSION CRITERIA:

* Average or maximum pain experienced greater than or equal to 50/100 on a visual analogue scale (average of data collected 7 days prior to the inclusion visit and recorded by the patient on the clinical diary)
* Evaluation by multidisciplinary team including neuro-surgeons, algologists and psychologists performed, (if not already done in the previous year for algologists and psychologists)
* Given informed consent.

EXCLUSION CRITERIA:

* Pregnant, or planning to become pregnant during the study (12months)
* Adults under guardianship or trusteeship
* Being treated or has been treated with spinal cord stimulation, subcutaneous or peripheral nerve stimulation, intrathecal drug delivery system.
* Had pudendal nerve decompression surgery less than 12 months ago
* Is suspected of substance abuse
* Has unresolved major issues of secondary gain
* Exhibits major psychiatric morbidity
* Has life expectancy inferior to 5 years
* Implant spinal cord stimulation surgery contraindication :

  * Magnetic resonnance imaging contraindication
  * History of coagulation disorder
  * Severe immunodepression, systemic, due to medicine drug intake or not (AIDS, transplanted, under anti TNF alpha treatment, …)
  * Current infection
* Would be unable to operate the spinal cord stimulation equipment, undergo the study assessments or complete questionnaires or clinical diary, based on the opinion of the investigator
* Unwilling to be treated with spinal cord stimulation, comply with study requirements.
* Suffering from another neuropathic pain, or chronic pain, cancer, diabetic neuropathy
* Patient with cardiac sentry stimulator or planned to be implanted with one

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Improvement of the sitting time from baseline to 6 months of follow-up | At 6 months of follow-up
  Sitting time is measured by a sitting time diary (in minutes) which patients will record during a daily activity, two times per day, once in the morning and once in the evening during one week before clinical visit.

SECONDARY OUTCOMES:
Improvement of the sitting time, as measured from baseline to 12 months of follow-up. | 12 months
  Sitting time is measured by a sitting time diary (in minutes) which patients will record during a daily activity, two times per day, once in the morning and once in the evening during one week before clinical visit.
Improvement of the sitting time, as measured from baseline to 3 months of follow-up. | 3 months
  Sitting time is measured by a sitting time diary (in minutes) which patients will record during a daily activity, two times per day, once in the morning and once in the evening during one week before clinical visit.
Improvement of the sitting time, as measured from baseline to 1 month of follow-up. | 1 month
  Sitting time is measured by a sitting time diary (in minutes) which patients will record during a daily activity, two times per day, once in the morning and once in the evening during one week before clinical visit.
Pain relief (visual analogic scale), as measured from baseline to 12 months of follow-up. | 12 months
  Visual analogic scale is recorded in a diary, which patient will complete two times per day, once in the morning and once in the evening during one week before clinical visit.
Pain relief (visual analogic scale), as measured from baseline to 6 months of follow-up. | 6 months
  Visual analogic scale is recorded in a diary, which patient will complete two times per day, once in the morning and once in the evening during one week before clinical visit.
Pain relief (visual analogic scale), as measured from baseline to 3 months of follow-up. | 3 months
  Visual analogic scale is recorded in a diary, which patient will complete two times per day, once in the morning and once in the evening during one week before clinical visit.
Pain relief (visual analogic scale), as measured from baseline to 1 month of follow-up. | 1 month
  Visual analogic scale is recorded in a diary, which patient will complete two times per day, once in the morning and once in the evening during one week before clinical visit.
Euro Quality of Life-5 Dimension Health questionnaire, as measured from baseline to 12 months of follow-up. | 12 months
  health-related quality of life
Use of pain treatment | 12 months
  Use of antiepileptics and of antidepressants and of analgesics OMS level I, II or III will be recorded and percentage of their variation between visits analysed.
  Use of non drugs therapies will be reported for descripton only.
Use of pain treatment | 6 months
  Use of antiepileptics and of antidepressants and of analgesics OMS level I, II or III will be recorded and percentage of their variation between visits analysed.
  Use of non drugs therapies will be reported for descripton only.
Use of pain treatment | 3 months
  Use of antiepileptics and of antidepressants and of analgesics OMS level I, II or III will be recorded and percentage of their variation between visits analysed.
  Use of non drugs therapies will be reported for descripton only.
Use of pain treatment | 1 month
  Use of antiepileptics and of antidepressants and of analgesics OMS level I, II or III will be recorded and percentage of their variation between visits analysed.
  Use of non drugs therapies will be reported for descripton only.
Euro Quality of Life-5 Dimension Health questionnaire, as measured from baseline to 6 months of follow-up | 6 months
  health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: BUFFENOIR Kevin, Professor, Principal Investigator — Nantes University Hospital
Locations (7):
- France (7):
  - Nantes Hospital, Nantes, Pays de la Loire Region
  - Bordeaux University Hospital, Bordeaux
  - Colmar Hospital, Colmar
  - Lille University Hospital, Lille
  - Lyon University Hospital, Lyon
  - Clinic Catherine de Sienne, Nantes
  - Hôpital Foch, Suresnes